CLINICAL TRIAL: NCT02854124
Title: Melanoma Cells Dissemination Study in Healthy Patients' Tissues
Brief Title: Tracing Dissemination of Melanoma Cells in Healthy Tissues
Acronym: DISSEMELA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI15020
Record Dates: First submitted 2016-07-31; First posted 2016-08-03 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Melanoma
Keywords: Melanoma; Dissemination; Initiating stem cells
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Primary melanoma, sentinel lymph node and peritumoral skin tissu
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with stage Ib and II melanoma: Melanoma and peritumoral skin excision
  Interventions: Procedure: Melanoma and peritumoral skin excision

INTERVENTIONS:
Procedure: Melanoma and peritumoral skin excision — Surgical retrieval of the primary tumor and safety retrieval of the surrounding normal peritumoral skin and sentinel lymph node

SUMMARY:
The objective of this project is to evaluate the presence of melanoma quiescent or initiating clonal cells in peritumoral healthy tissue displaying the same molecular signature than those of the tumor/metastasis and to correlate this presence to the prognostic value.

DETAILED DESCRIPTION:
In the western world, melanoma incidence has constantly risen for the last 50 years, and it is currently reported as the most frequent tumor in 20 - 29 year old women. BRAF, NRAS and c-kit genes play an important role in cell proliferation and are mutated at very high frequency in melanoma. Despite the recent therapeutical breakthroughs obtained with the use of new drugs, metastatic melanoma remains still a life threatening disease. One of the main questions in melanoma concern the initial steps leading to metastatic spread, a better understanding being a key step to its prevention and the identification of new molecular mechanisms being implemental to the improvement of our therapeutical arsenal.

The proposed work aims to study the hypothesis of early spread in human melanoma using the recently developed powerful techniques of e-ice cold PCR, as well as classical immunohistochemistry. To do so, investigators will take advantage on the fact that treatment of melanoma relies on a secondary excision of normal peritumoral skin and sentinel lymph node. This peritumoral tissue is large (measuring 2 to 6 cm diameter), contains lymphatics in the hypodermis, the tissue considered to host the metastatic route of melanocytes and remains partially available for analysis.

All patients with stage Ib and II melanoma followed in the parisian cohort Melan-cohort, Cochin Hospital and Gustave Roussy Institute included between 2005 and 2009 will be found. A PCR analysis will be done on DNA extracted from paraffin embedded sections of primary tumors. Patients who display mutations in BRAF (BRAFV600E, BRAFV600K), NRAS (codon 61) or c-kit genes will be selected. The archival paraffin embedded tissues from healthy perilesional skin as well as from healthy sentinel lymph nodes will be obtained. Pyrosequencing and e-ice cold PCR targeting the mutations of the above genes at their usual positions will be done on DNA extracted from these specimens. Immunofluorescence anti-BRAFV600E or anti tumoral/initiating/stem cells will be done on same tissues. These simple techniques will test -using a sensitive molecular biology tool- whether in humans with melanomas, there is early dissemination of melanoma cells in histopathological healthy sentinel lymph node and peritumoral skin. The presence of these clonal cells in these healthy tissues will be correlated to the survival of the patients after 5 years and will allow the development of new therapeutic follow-up and strategies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age > 18 years old.
* Primary melanomas stage Ib and II.
* Melanomas mutated BRAF, NRAS, c-kit.
* Cutaneous melanomas.

Exclusion Criteria:

* Metastatic melanomas stage III and IV.
* Melanomas with invasion of the peritumoral skin tissue.
* Congenital or acquired immunosuppression.
* Antitumoral, immunosuppressive treatments or any other diseases during the follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage Ib and II melanoma followed in the parisian cohort Melan-cohort, Cochin Hospital and Gustave Roussy Institute included between 2005 and 2009
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Survival at 5 years | 5 years
  correlation to the presence of tumoral initiating stem cells in healthy tissues

SECONDARY OUTCOMES:
Survival at 5 years without tumor recurrence | 5 years
  correlation to the presence of tumoral initiating stem cells in healthy tissues

CONTACTS AND LOCATIONS:
Overall Officials: Romain Fontaine, PhD, Principal Investigator — INSERM - UMRS 938
Locations (1):
- Name:: INSERM - UMRS 938, UPMC Saint-Antoinen Hospital, Team "Stem cells and transition from pre-invasive tumors", Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curtin JA, Fridlyand J, Kageshita T, Patel HN, Busam KJ, Kutzner H, Cho KH, Aiba S, Brocker EB, LeBoit PE, Pinkel D, Bastian BC. Distinct sets of genetic alterations in melanoma. N Engl J Med. 2005 Nov 17;353(20):2135-47. doi: 10.1056/NEJMoa050092. PMID 16291983
- [Background] Faries MB, Steen S, Ye X, Sim M, Morton DL. Late recurrence in melanoma: clinical implications of lost dormancy. J Am Coll Surg. 2013 Jul;217(1):27-34; discussion 34-6. doi: 10.1016/j.jamcollsurg.2013.03.007. Epub 2013 May 3. PMID 23643694
- [Background] Quintana E, Shackleton M, Sabel MS, Fullen DR, Johnson TM, Morrison SJ. Efficient tumour formation by single human melanoma cells. Nature. 2008 Dec 4;456(7222):593-8. doi: 10.1038/nature07567. PMID 19052619
- [Background] How-Kit A, Tost J. Pyrosequencing(R)-Based Identification of Low-Frequency Mutations Enriched Through Enhanced-ice-COLD-PCR. Methods Mol Biol. 2015;1315:83-101. doi: 10.1007/978-1-4939-2715-9_7. PMID 26103893